CLINICAL TRIAL: NCT03081260
Title: Long-term Evaluation Protocol (12 Months Postoperative) of Total Knee Prostheses Anatomic With Resurfaced Patella Versus Non-resurfaced Patella in Patients Requiring Total Knee Arthroplasty Prospective, Monocentric, Randomized, Open-label Study
Brief Title: Long-term Evaluation Protocol (12 Months Postoperative) of Total Knee Prostheses Anatomic With Resurfaced Patella Versus Non-resurfaced Patella in Patients Requiring Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL16_0645; 2016-A01697-44 (Other: ANSM)
Record Dates: First submitted 2017-03-09; First posted 2017-03-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Arthroplasty
Keywords: Total Knee Arthroplasty; Patella; Resurfacing; IKS score
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patellar resurfacing (Other): Patellar resurfacing during the total knee prosthesis Anatomic surgery
  Interventions: Other: Patellar resurfacing
- Patellar non-resurfacing (Other): Patellar non-resurfacing during the total knee prosthesis Anatomic surgery
  Interventions: Other: Patellar non-resurfacing

INTERVENTIONS:
Other: Patellar resurfacing — The resurfacing of the patella is generally done at the end of the surgery, after having ejected the patella. A frontal bone cut is made using a dedicated ancillary to remove the entire cartilage. Orifices are then made in the patella so that the polyethylene implant can be accommodated with studs which will be cemented on the joint face of the ball joint.
  Arms: Patellar resurfacing
Other: Patellar non-resurfacing — Non-resurfacing of the patella does not involve any additional surgical action
  Arms: Patellar non-resurfacing

SUMMARY:
Total knee arthroplasty is a frequent surgery in France. It currently represents 70,000 interventions per year. The total knee prosthesis is also called tri-compartmental because it allows articulation between the femur and the tibia but also between the femur and the patella.

The patella belongs to the extensor system. It articulates with the femoral trochlea in which it slides. It has an important biomechanical role on the quadriceps strength in addition to allowing flexion-extension movements.

In the case of resurfacing, the joint face of the patella is cut off; A convex polyethylene implant is sealed with cement using studs on the same face.

In case of non-resurfacing, the surgeon leaves in place the cartilage of the patella which will be in direct contact with the femoral prosthetic trochlea.

Both methods have advantages and disadvantages. For some implants, it is recommended to resurface the patella because the implant is not very tolerant with the native patella. Other implants have been designed to be better adapted to the preservation of patellar cartilage.

There is currently no evidence that one method is superior to the other on new generation implants known as "patellar friendly".

It seems necessary to compare both methods in terms of long-term postsurgery results.

DETAILED DESCRIPTION:
The analysis of the primary endpoint (International Knee Society score (IKS score)) will be based on the assumption that the postsurgery score will be identical in both groups. The t test for independent samples will be used to test this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female (age ≥ 18 years)
* Diagnosis of knee arthrosis (internal femoro-tibial arthrosis, external femorotibial osteoarthritis, femoro-patellar arthrosis)
* Indication of total first-line knee arthroplasty

Exclusion Criteria:

* Patient whose surgical complexity requires the placement of a strained prosthesis (ligament laxity, bone loss).
* Refusal to participate in the study
* Pregnant women, parturients or nursing mothers
* Persons deprived of their liberty by a judicial or administrative decision, persons subject to psychiatric care, persons admitted to a health or social institution for purposes other than research
* Minor Patients
* Major persons who are subject to a legal protection measure or are unable to express their consent
* Patient not affiliated to a social security scheme
* Patient participating in other interventional research excluding routine care studies not interfering with analysis of primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
measure of International Knee Society score (IKS score) | 12 months after surgery
  The comparison of the IKS (International Knee Society) scores (2011 version) will be done between both groups.

SECONDARY OUTCOMES:
abnormality of the patellar stroke | 12 months after surgery
  Presence of an abnormality of the patellar stroke with the type of tilting, subluxation or dislocation of the patella on the X-ray images.
Measure of the forgotten joint score | 12 months after surgery
  The comparison of the forgotten joint score will be done between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Lustig, MD, Principal Investigator — Hôpital de la Croix-Rousse
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Deroche E, Batailler C, Swan J, Sappey-Marinier E, Neyret P, Servien E, Lustig S. No difference between resurfaced and non-resurfaced patellae with a modern prosthesis design: a prospective randomized study of 250 total knee arthroplasties. Knee Surg Sports Traumatol Arthrosc. 2022 Mar;30(3):1025-1038. doi: 10.1007/s00167-021-06521-y. Epub 2021 Mar 4. PMID 33661323